CLINICAL TRIAL: NCT05577975
Title: Pilot Evaluation of Technology-enhanced Horticultural Activities Among the People With Dementia and Their Family Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Patrick KOR Pui Kin, Assistant Professor, School of Nursing, The Hong Kong Polytechnic University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSEARS20220801002
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): The program will consist of three face-to-face (F-T-F) horticultural activity training session for a group of 6-8 participants and then biweekly telephone follow-up for 8-week home-based horticultural intervention.
  Interventions: Device: The Aspara @ smart grower

INTERVENTIONS:
Device: The Aspara @ smart grower — The program will consist of three face-to-face (F-T-F) horticultural activity training session for a group of 6-8 participants and then biweekly telephone follow-up for 8-week home-based horticultural intervention. The home-based program contains different horticultural, cognitive and multisensory stimulation activities such asking the PWD and the family caregiver to record the sense of touch and odor when taking care of the plant and the various changes of the plants by using the smart grower. Program evaluation will be conducted through focus groups with 15 participants with different levels of stress reduction after the intervention.

SUMMARY:
Horticultural therapy is one of the effective interventions for the person with dementia(PWD) which could increase their time engaging in leisure activities and decrease their time doing nothing. However, there are some limitations and constraints for PWD to participate in the horticultural therapy especially in the high-density cities (e.g. Hong Kong). This study aims to investigate the feasibility and preliminary effects of adopting home-based technology-enhanced horticultural activities. The program will consist of three face-to-face (F-T-F) horticultural activity training session for a group of 6-8 participants and then biweekly telephone follow-up for 8-week home-based horticultural intervention. Program evaluation will be conducted through focus groups with 15 participants with different levels of stress reduction after the intervention. It is hypothesized that the PWD and their caregiver will have a significant improvement in the cognitive function and behavioral symptoms of the PWD, an increase in the positive caregiving experience in the family caregivers, a reduction of the caregivers' level of stress and depressive symptoms, and enhancement of the quality of life of the family caregivers after the intervention.

DETAILED DESCRIPTION:
Objective This study aims to investigate the feasibility and preliminary effects of adopting home-based technology-enhanced horticultural activities to: a) improve the cognitive function and behavioral symptoms of the PWD; b) promote the positive caregiving experience in the family caregivers; c) reduce the caregivers' level of stress and depressive symptoms; and d) improve the quality of life of the family caregivers. To the best of our knowledge, it is the first program adopting Smart Grower for horticultural intervention among the PWD and their family caregivers in Hong Kong.

Method The home-based technology-enhanced horticultural activities will be delivered for the people with dementia and their family caregivers through a smart grower. The smart grower is a hydroponic indoor grower that builds a controllable environment with auto optimization for growing healthy plants, fresh vegetables, herbs, and fruits. A mobile app will be connected to the grower for controlling the growing environment (e.g. lighting, watering), tracking the progress of the plants, guiding the older people with dementia and their family caregiver to conduct the horticulture activities. The program will consist of three face-to-face (F-T-F) horticultural activity training session for a group of 6-8 participants and then biweekly telephone follow-up for 8-week home-based horticultural intervention. The home-based program contains different horticultural, cognitive and multisensory stimulation activities such asking the PWD and the family caregiver to record the sense of touch and odor when taking care of the plant and the various changes of the plants by using the smart grower. Program evaluation will be conducted through focus groups with 15 participants with different levels of stress reduction after the intervention. The aims of the focus groups is to identify the strengths, limitations, and difficulties of the home-based technology-enhanced horticultural program.

Significance and Value In this project, we would like to collaborate with the elderly center to deliver the technology-enhanced horticultural activities for PWD in the community and make this program sustainable in the community. Meanwhile, we will collect the users' feedback and further modify the program to fit the needs of the people with dementia and the family caregivers.

In the future, we hope that the program will not only benefit the community-dwelling older people but also those receiving service in the respite center, day care center, hospice and nursing home as they are also facing the challenges of manpower shortage, issues of loneness and poor psychological health. We will base on the data and results collected from this proposed study and further revise the program and software for servicing the older people in nursing through a group-based approach.

ELIGIBILITY:
Inclusion Criteria:

1. The PWD

   1. Aged 65 or above who had been diagnosed with any type of dementia at the early to moderate stage
   2. Are Community-dwelling (i.e., non-institutionalized),
   3. Are Able to understand Cantonese and follow simple instruction
2. The family caregivers

   1. Aged 18 years or above;
   2. the blood or by-marriage relatives (e.g. spouses, siblings, children, and grandchildren) of a person who has been clinically diagnosed with dementia, regardless of its types and these relatives are taking up the caring responsibilities ranging from physical aids to emotional supports, in the form of transportation, financial assistance, personal hygiene, and decision-making.;
   3. Providing most of the daily care and support for PWD (daily contact for at least four hours); and
   4. Able to speak Cantonese

Exclusion Criteria:

The PWD and the family caregivers

1. Are diagnosed with a mental disorder such as bipolar disorder, schizophrenia, dementia, or depression; and/or,
2. Are taking anticonvulsants, or any kind of psychotropic drugs, and/or identified with a self-reported suicidal thought or drug abuse in the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
The Chinese version of Positive Aspect of Caregiving scale (PAC) | At baseline (T0) and 11th week (immediately post- intervention; T1
  The PAC scale demonstrates the acceptable levels of internal consistency Cronbach's alpha 0.85 among the family caregivers of PWD in Hong Kong. Higher scores indicating more positive self-perceptions of caregiving. Comparisons of changes of Positive Aspect of Caregiving scale (PAC)will be considered as follows: T0 - T1
The Chinese version of Perceived Stress Scale (PSS) | At baseline (T0) and 11th week (immediately post- intervention; T1
  Perceived Stress Scale contains 10 items with 5-point Likert-type scale rating from 0 (never) to 4 (very often). The total score can range from 0 to 40 with higher scores indicating higher perceived stress. Comparisons of changes of Perceived Stress Scale will be considered as follows: T0 - T1
The WHOQOL-OLD BREF (HK) | At baseline (T0) and 11th week (immediately post- intervention; T1
  The WHOQOL-OLD BREF (HK) comprised 28 items and each item is rated on a 5-point Likert-type scale that ranged from 1 (very dissatisfied) to 5 (very satisfied), with a higher score indicating a better QoL. Comparisons of changes of The WHOQOL-OLD BREF (HK) will be considered as follows: T0 - T1
The Chinese version of Center for Epidemiological Studies Depression scale(CESDS) | At baseline (T0) and 11th week (immediately post- intervention; T1
  The Chinese version of Center for Epidemiological Studies Depression scale is a self-reported measure of depression containing 20 items. Comparisons of changes of Center for Epidemiological Studies Depression scale will be considered as follows: T0 - T1
MoCA-5-min | At baseline (T0) and 11th week (immediately post- intervention; T1
  MoCA-5-min assess participants' cognitive function over the telephone. MoCA-5-min comprises four domains: attention, executive function/language, orientation, and memory.Comparisons of changes of MoCA-5-min will be considered as follows: T0 - T1
The Chinese version of the Neuropsychiatric Inventory-Questionnaire (NPI-Q) | At baseline (T0) and 11th week (immediately post- intervention; T1
  The Neuropsychiatric Inventory-Questionnaire evaluates the frequency, severity, and caregiver distress of 12 neuropsychiatric symptoms by using a 5-point rating scale..Comparisons of changes of the Neuropsychiatric Inventory-Questionnaire will be considered as follows: T0 - T1

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kor, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic Univeristy, Hong Kong, Hong Kong

REFERENCES:
- [Background] Chau, P. H., McGhee, S. M., Yu, R., Cheung, W. L., Chan, K. C., Cheung, S. H., & Woo, J. (2010). Dementia Trends: Impact of the Ageing Population and Societal Implications for Hong Kong. Hong Kong: The Hong Kong Jockey Club.
- [Background] Chin WY, Choi EP, Chan KT, Wong CK. The Psychometric Properties of the Center for Epidemiologic Studies Depression Scale in Chinese Primary Care Patients: Factor Structure, Construct Validity, Reliability, Sensitivity and Responsiveness. PLoS One. 2015 Aug 7;10(8):e0135131. doi: 10.1371/journal.pone.0135131. eCollection 2015. PMID 26252739
- [Background] Chu, L. C., & Kao, H. S. (2005). The moderation of meditation experience and emotional intelligence on the relationship between perceived stress and negative mental health (Vol. 47).
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Laver K, Milte R, Dyer S, Crotty M. A Systematic Review and Meta-Analysis Comparing Carer Focused and Dyadic Multicomponent Interventions for Carers of People With Dementia. J Aging Health. 2017 Dec;29(8):1308-1349. doi: 10.1177/0898264316660414. Epub 2016 Jul 25. PMID 27458254
- [Background] Leung DY, Lam TH, Chan SS. Three versions of Perceived Stress Scale: validation in a sample of Chinese cardiac patients who smoke. BMC Public Health. 2010 Aug 25;10:513. doi: 10.1186/1471-2458-10-513. PMID 20735860
- [Background] Lin Y, Lin R, Liu W, Wu W. Effectiveness of horticultural therapy on physical functioning and psychological health outcomes for older adults: A systematic review and meta-analysis. J Clin Nurs. 2022 Aug;31(15-16):2087-2099. doi: 10.1111/jocn.16095. Epub 2021 Oct 24. PMID 34694042
- [Background] Lou VW, Lau BH, Cheung KS. Positive aspects of caregiving (PAC): scale validation among Chinese dementia caregivers (CG). Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):299-306. doi: 10.1016/j.archger.2014.10.019. Epub 2014 Nov 7. PMID 25488014
- [Background] Lu LC, Lan SH, Hsieh YP, Yen YY, Chen JC, Lan SJ. Horticultural Therapy in Patients With Dementia: A Systematic Review and Meta-Analysis. Am J Alzheimers Dis Other Demen. 2020 Jan-Dec;35:1533317519883498. doi: 10.1177/1533317519883498. Epub 2019 Nov 5. PMID 31690084
- [Background] Ng KST, Sia A, Ng MKW, Tan CTY, Chan HY, Tan CH, Rawtaer I, Feng L, Mahendran R, Larbi A, Kua EH, Ho RCM. Effects of Horticultural Therapy on Asian Older Adults: A Randomized Controlled Trial. Int J Environ Res Public Health. 2018 Aug 9;15(8):1705. doi: 10.3390/ijerph15081705. PMID 30096932
- [Background] Prince M, Bryce R, Albanese E, Wimo A, Ribeiro W, Ferri CP. The global prevalence of dementia: a systematic review and metaanalysis. Alzheimers Dement. 2013 Jan;9(1):63-75.e2. doi: 10.1016/j.jalz.2012.11.007. PMID 23305823
- [Background] Radloff, L. S. (1977). The CES-D scale: A self-report depression scale for research in the general population. Applied psychological measurement, 1(3), 385-401.
- [Background] Van't Leven N, Prick AE, Groenewoud JG, Roelofs PD, de Lange J, Pot AM. Dyadic interventions for community-dwelling people with dementia and their family caregivers: a systematic review. Int Psychogeriatr. 2013 Oct;25(10):1581-603. doi: 10.1017/S1041610213000860. Epub 2013 Jul 24. PMID 23883489
- [Background] Wong A, Cheng ST, Lo ES, Kwan PW, Law LS, Chan AY, Wong LK, Mok V. Validity and reliability of the neuropsychiatric inventory questionnaire version in patients with stroke or transient ischemic attack having cognitive impairment. J Geriatr Psychiatry Neurol. 2014 Dec;27(4):247-52. doi: 10.1177/0891988714532017. Epub 2014 Apr 24. PMID 24763069
- [Background] Wong A, Nyenhuis D, Black SE, Law LS, Lo ES, Kwan PW, Au L, Chan AY, Wong LK, Nasreddine Z, Mok V. Montreal Cognitive Assessment 5-minute protocol is a brief, valid, reliable, and feasible cognitive screen for telephone administration. Stroke. 2015 Apr;46(4):1059-64. doi: 10.1161/STROKEAHA.114.007253. Epub 2015 Feb 19. PMID 25700290
- [Background] Wong A, Xiong YY, Kwan PW, Chan AY, Lam WW, Wang K, Chu WC, Nyenhuis DL, Nasreddine Z, Wong LK, Mok VC. The validity, reliability and clinical utility of the Hong Kong Montreal Cognitive Assessment (HK-MoCA) in patients with cerebral small vessel disease. Dement Geriatr Cogn Disord. 2009;28(1):81-7. doi: 10.1159/000232589. Epub 2009 Aug 11. PMID 19672065
- [Background] Yu R, Chau PH, McGhee SM, Cheung WL, Chan KC, Cheung SH, Woo J. Trends in prevalence and mortality of dementia in elderly Hong Kong population: projections, disease burden, and implications for long-term care. Int J Alzheimers Dis. 2012;2012:406852. doi: 10.1155/2012/406852. Epub 2012 Oct 14. PMID 23097740
- [Background] Zhao Y, Liu Y, Wang Z. Effectiveness of horticultural therapy in people with dementia: A quantitative systematic review. J Clin Nurs. 2022 Jul;31(13-14):1983-1997. doi: 10.1111/jocn.15204. Epub 2020 Feb 20. PMID 32017241
- [Derived] Kor PPK, Liu JYW, Wong AKC, Tsang APL, Tan HZ, Cheung DSK, Leung HKW, Wong FKY. Effectiveness of a Dyadic Technology-Enhanced Home-Based Horticultural Therapy on Psychosocial Well-Being Among People With Dementia and Their Family Caregivers: Multimethods Pilot Study. JMIR Aging. 2025 Feb 5;8:e66017. doi: 10.2196/66017. PMID 39908077